CLINICAL TRIAL: NCT04407728
Title: Early Detection of Severe Heart Disease in Fetuses at High Risk of Heart
Brief Title: Early Detection of Severe Heart Disease in Fetuses at High Risk of Heart Disease
Acronym: PRECAFOET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC20.009
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- precocious EchoMorpho-T1 (Experimental): Women whose fetus is at high risk of congenital heart disease after the 1st trimester screening echo (EchoT1), will benefit from an early morphological ultrasound centered on the heart (EchoMorpho-T1) by a sonographer referent between 11 and 14 weeks +/- of an early fetal heart ultrasound (EchoCoeur-T1) between 11 and 15 weeks by a cardio-pediatrician in the event of an abnormality with the EchoMorpho-T1.
  Interventions: Other: early ultrasound screening

INTERVENTIONS:
Other: early ultrasound screening — Women whose fetus is at high risk of congenital heart disease at the end of the 1st trimester screening ultrasound (EchoT1), will benefit from an early heart-centered morphological ultrasound (EchoMorpho-T1) by a referring sonographer between 11 and 14 SA +/- an early fetal cardiac ultrasound (EchoCoeur-T1) between 11 and 15 SA by a cardio-paediatrician in case of EchoMorpho-T1 abnormality.
  The results of the early morphological and cardiac ultrasounds will be compared with those of the 2nd trimester ultrasound at 18-22SA (EchoMorpho-T2) and +/- of the fetal cardiac ultrasound between 18SA and 24SA (Gold standard) or, failing this, with the anatomopathological examination when it is available if a medical termination of pregnancy took place before the EchoMorpho-T2.

SUMMARY:
The main objective of the work is to evaluate, in the French health care system, the performance of early ultrasound screening for severe heart disease between 11 and 14SA in high-risk populations.

DETAILED DESCRIPTION:
Numerous studies have shown a link between increased nuchal translucency and heart disease. Although high-risk fetal populations are identified between 11 and 13 SA on clinical and biological criteria and by screening ultrasound (Echo T1), cardiac morphology analysis is routinely performed only during 2nd trimester fetal morphology ultrasound between 18 and 22 SA (EchoMorpho-T2) inducing a difficult wait for the couple.

The development of increasingly efficient ultrasound probes has made it possible to explore the foetal heart at an earlier stage. International learned societies recommend an early morphological examination with heart-centered slices before 14 weeks in high-risk situations. This practice is not systematic in France and no study has evaluated its feasibility and impact in a French care network.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women whose fetus is at high risk for congenital heart disease:

* Nuchal translucency measurement on T1 echo ≥3.5mm
* Cardiac or extra-cardiac morphological abnormality suspected on the T1 screening echo
* First degree family history for the fetus (patient, spouse, 1st children of the couple) of significant congenital cardiopathy (excluding AIC, muscular VIC or persistent CA).

Exclusion Criteria:

* Multiple Pregnancies
* non-emancipated minors, persons unable to express their consent.
* Lack of affiliation to a social security scheme.
* Subject in a period of exclusion from another study,
* Subject under administrative or judicial supervision
* Subject cannot be contacted in case of emergency

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2022-05-02 (Estimated); Study Completion 2022-11-02 (Estimated)

PRIMARY OUTCOMES:
early ultrasound screening | 1 day
  Calculation of the sensitivity and specificity of screening for severe heart disease using EchoMorpho-T1. Specificity will be privileged in order to avoid the anxiety-producing nature of false positives.

IPD SHARING:
Plan to Share IPD: Undecided